CLINICAL TRIAL: NCT05237102
Title: Prediction Model of Improvement of Disturbance of Consciousness in Patients With Hydrocephalus After Shunt Operation: Based on Patient Preoperative Imaging, EEG and Lumbar Tap Test
Brief Title: Prediction Model of Improvement of Disturbance of Consciousness in Patients With Hydrocephalus After Shunt Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhuohang Wang (Other)
Responsible Party: Sponsor-Investigator, Zhuohang Wang, Principal Investigator, Nanchang University
Organization: Nanchang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: NanchangUZWang
Record Dates: First submitted 2021-12-16; First posted 2022-02-11 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Disorder of Consciousness; Hydrocephalus
Keywords: shunt; tap test
MeSH Terms: conditions — Consciousness Disorders; Hydrocephalus | interventions — Cerebrospinal Fluid Shunts

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The patients did not respond to CSF tap test (Experimental): Participants assigned to the experimental group did not respond to the CSF tap test and did not show improvement in general symptoms of hydrocephalus and disturbance of consciousness, but there may be changes in eeg and imaging parameters (it is unknown whether such changes are related to surgical outcome).
  Interventions: Procedure: Cerebrospinal fluid shunt
- The patients did respond to CSF tap test (Other): The improvement of symptoms in these participants after the CSF tap test predicts a favorable prognosis for CSF shunt.
  Interventions: Procedure: Cerebrospinal fluid shunt

INTERVENTIONS:
Procedure: Cerebrospinal fluid shunt — The procedure is designed to reduce the amount of cerebrospinal fluid in a patient's brain by draining it through a shunt tube:
  ①V-P shunt is suitable for most types of hydrocephalus; ②L-P shunt is suitable for traffic hydrocephalus and positive pressure hydrocephalus, and patients with lower cerebellar tonsil hernia are contraindications; ③ Common terms of ventriculoatrial (V-A) shunt are not suitable for V-P shunt (abdominal infection, serious respiratory and circulatory diseases are contraindications); ④ The third ventriculostomy is suitable for patients with non-traffic and partial traffic hydrocephalus （infants and patients with severe ventricular enlargement should be cautious, and patients with shunt tube cannot be placed due to ventricular conditions）; ⑤Other shunt methods include septum pellucidum fistula and Torshunt （ventriculo-occipital cistern shunt after tumor resection）

SUMMARY:
Patients with hydrocephalus are usually treated with cerebrospinal fluid (CFS) shunt to deal with excess cerebrospinal fluid in the brain. However, it is difficult to distinguish whether ventricular enlargement is due to hydrocephalus or other causes, such as brain injury and compensatory brain atrophy after surgery. Therefore, it is important to predict whether shunting will help patients. For this reason, clinicians must be cautious when treating patients with shunt therapy. Important assessments of the level of consciousness and continuous lumbar tap test are currently clinically common predictors before making decisions about CFS shunt therapy. However, for patients with serious disturbance of consciousness, it is difficult to predict the prognosis of surgery by observing the improvement of symptoms after lumbar tap test, which brings difficulties to the majority of clinical workers, and also easy to bring serious psychological and economic burden to patients.

In clinical practice, clinicians still lack a stable and objective method to predict postoperative outcomes for these patients.

In this clinical study, when participants performed the cerebrospinal fluid tap test to evaluate whether or not cerebrospinal fluid shunt was performed, various predictors that may be associated with CSF shunt outcomes before and after cerebrospinal fluid tap test were collected, including imaging data, EEG characteristics and changes in cerebrospinal fluid pressure. In addition, the researchers will collect the improvement of consciousness disturbance in patients with hydrocephalus before and after cerebrospinal fluid shunt, in order to explore the correlation between preoperative imaging data, EEG characteristics, the results of cerebrospinal fluid tap test and the improvement of consciousness disorders. A scheme of consciousness assessment based on the results of imaging, EEG and tap test results afte CSF tap test was proposed.

DETAILED DESCRIPTION:
Among them, imaging parameters include:

Evans index, EI; Callosal angle, CA; Z-Evans index, Z-EI; Brain/ventricle ratio, BVR; Frontal horn ratio, FHR; Frontal and occipital horn ratio, FOR/FOHR; Frontal and Temporal Horn Ratio, FTHR; Bicaudate ratio，BCR; Cella media ratio, CMR, etc. and the disorder of consciousness scales include: Coma recovery scale-Revised，CRS-R Glasgow-Pittsburgh cerebral performance categories Glasgow coma scale, GCS, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, gender is not limited.
* Patients with traffic hydrocephalus caused by various reasons, including atmospheric hydrocephalus, who need cerebrospinal fluid shunt and meet the surgical indications to a certain extent.
* Typical imaging manifestations of hydrocephalus patients.
* Clinical manifestations of consciousness disorder.
* Whether or not you can participate in the study will be decided after a doctor's examination.

Exclusion Criteria:

* patients with mental or motor disorders, such as Alzheimer's disease, schizophrenia, and Parkinson's disease.
* Patients with abnormal coagulation mechanism or receiving treatment with thrombolysis agent, anticoagulant or platelet coagulant inhibitor and hemophilia.
* Patients with serious diseases of other systems, such as serious diseases of blood system, respiratory system, digestive system, urinary system and immune system, as well as patients with mental disorders and recent history of intracranial infection.
* Patients with a known disease causing ventricle enlargement.
* Female patients in pregnancy and lactation.
* Other circumstances in which the doctor judges that he cannot participate in the test.
* The subject himself or his legal representative refuses to participate in the clinical trial. Whether you are suitable to participate in this study needs the final decision after doctor's examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Changes of consciousness disorder after operation | 24 hours after surgery
  The score of the scale Coma recovery scale-Revised will be used to assess changes in consciousness before and after surgery (the highest score is 23 points and the lowest score is 0 points. A higher score indicates a better prognosis)
Changes of consciousness disorder after operation | 14 days after surgery
  The score of the scale Coma recovery scale-Revised will be used to assess changes in consciousness before and after surgery (the highest score is 23 points and the lowest score is 0 points. A higher score indicates a better prognosis)
Changes of consciousness disorder after operation | 1 month after surgery
  The score of the scale Coma recovery scale-Revised will be used to assess changes in consciousness before and after surgery (the highest score is 23 points and the lowest score is 0 points. A higher score indicates a better prognosis)
Changes of consciousness disorder after operation | 6 months after surgery
  The score of the scale Coma recovery scale-Revised will be used to assess changes in consciousness before and after surgery (the highest score is 23 points and the lowest score is 0 points. A higher score indicates a better prognosis)

CONTACTS AND LOCATIONS:
Overall Officials: Xiangrong Wang, bachelor, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical trial had a separate Case Report Form customized for each participant, including the basic situation, state of the illness and prognosis of the patient. And the Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, Analytic Code are to be shared with other researchers too.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the completion of the trial to the completion of three years.
Access Criteria: NO/NA

REFERENCES:
- [Result] Arnts H, van Erp WS, Sanz LRD, Lavrijsen JCM, Schuurman R, Laureys S, Vandertop WP, van den Munckhof P. The Dilemma of Hydrocephalus in Prolonged Disorders of Consciousness. J Neurotrauma. 2020 Oct 15;37(20):2150-2156. doi: 10.1089/neu.2020.7129. Epub 2020 Jul 22. PMID 32484029
- [Result] Ozgode Yigin B, Algin O, Saygili G. Comparison of morphometric parameters in prediction of hydrocephalus using random forests. Comput Biol Med. 2020 Jan;116:103547. doi: 10.1016/j.compbiomed.2019.103547. Epub 2019 Nov 20. PMID 32001008
- [Result] Nakajima M, Yamada S, Miyajima M, Ishii K, Kuriyama N, Kazui H, Kanemoto H, Suehiro T, Yoshiyama K, Kameda M, Kajimoto Y, Mase M, Murai H, Kita D, Kimura T, Samejima N, Tokuda T, Kaijima M, Akiba C, Kawamura K, Atsuchi M, Hirata Y, Matsumae M, Sasaki M, Yamashita F, Aoki S, Irie R, Miyake H, Kato T, Mori E, Ishikawa M, Date I, Arai H; research committee of idiopathic normal pressure hydrocephalus. Guidelines for Management of Idiopathic Normal Pressure Hydrocephalus (Third Edition): Endorsed by the Japanese Society of Normal Pressure Hydrocephalus. Neurol Med Chir (Tokyo). 2021 Feb 15;61(2):63-97. doi: 10.2176/nmc.st.2020-0292. Epub 2021 Jan 15. PMID 33455998